CLINICAL TRIAL: NCT04082130
Title: Clinical Comparison of Coronally-advanced Flap Plus Xenogeneic Collagen Matrix (Fibro-Gide®) and Subepithelial Connective Tissue Graft in the Treatment of Gingival Recessions
Brief Title: Xenogenic Collagen Matrix and Subepithelial Connective Tissue Graft in the Treatment of Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Perio-01-2019
Record Dates: First submitted 2019-08-28; First posted 2019-09-09 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Gingival Recession Localized Moderate
Keywords: Xenogenic collagen matrix (XCM).; subepithelial connective tissue graft (SCGT).; coronally advanced flap (CAF).; Root coverage.

STUDY DESIGN:
Intervention Model Description: split-mouth design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (XCM)+(CAF) (Experimental): Surgical protocol for test treatment with CAF + XCM:
  After local anesthetizing the recipient site,CAF elevation will be done using (De Sanctis & Zucchelli 2007) design.Horizontal incisions will be done at the recession site,another two slightly divergent vertical incisions will be done at the end of previous incisions extending to the mucogingival junction.The resulting flap will be split thickness in the surgical papillae area,then will be full thickness exposing 3-4 mm of the bone apically of the dehiscence and after that it will be split thickness in the apical direction,all the muscle insertions will be eliminated,the root surface will be prepared by curettes and chemically treated with 24% EDTA gel.De-epithelialization of the interdental papillae will be done.The XCM will be trimmed and fix onto the root surface 1-2mm coronally of the CEJ using absorbable sutures,and the flap will be coronally advanced to fully cover the XCM and then sutured to the de-epithelialized papillae.
  Interventions: Procedure: (XCM)+(CAF)
- (SCTG)+(CAF) (Active Comparator): The surgical protocol in the control group will be identical with test group protocol with these exceptions:
  1. The entire flap will be elevated as split thickness instead of split-full-split thickness flap.
  2. A SCTG harvested from the palate will be used to cover the exposed denuded root surface in lieu of placement of XCM in the test group. And absorbable sutures will be used to stabilize it 2 mm coronally from the CEJ.
  3. As in the test group the mucosal flap will coronally advanced to completely cover the SCTG then sutured to the de-epithelialized papillae.
  Interventions: Procedure: (SCTG)+(CAF)

INTERVENTIONS:
Procedure: (XCM)+(CAF) — The description of this intervention has been already given before.
  Arms: (XCM)+(CAF)
Procedure: (SCTG)+(CAF) — The description of this intervention has been already given before.
  Arms: (SCTG)+(CAF)

SUMMARY:
this study is a Clinical evaluation of using Xenogenic collagen matrix (XCM) plus coronally advanced flap (CAF) compared to subepithelial connective tissue graft (SCTG) plus coronally advanced flap to treat Miller class I gingival recession. A split-full-split thickness flap will be elevated in the (XCM+CAF) group while it will be an only partial thickness flap in the (SCTG+CAF) group. The sample size will be 15 patients. Each patient has bilateral Miller Class I gingival recessions; and as a split-mouth study design one side will be treated with (SCTG+CAF), while the other will be treated with (XCM+CAF).

DETAILED DESCRIPTION:
The aim of this study is to clinically compare between the subepithelial connective tissue graft (SCTG) plus coronally advanced flap (CAF) which is defined as the golden standard for the treatment of gingival recessions and Xenogenic collagen matrix (XCM) plus coronally advanced flap (CAF) to treat class I Miller gingival recession. CAF elevation will be done as it described by (De Sanctis & Zucchelli 2007) with modifications in the the control group.The flap will be partially elevated in the (SCTG+CAF) group while it will be a split-full-split thickness flap in the (XCM+CAF) group, and finally the flap will stabilized coronally. Fifteen patients who have bilateral buccal Miller Class I gingival recession defects will be enrolled in this study. These defects will be distributed randomly into two groups: the test group (XCM+CAF) and control group (SCTG+CAF). Clinical parameters will be evaluated: Recession depth (REC), change in visible plaque index, recession width (RW), width of keratinized tissue (KT), thickness of gingival tissue (GT), probing depth (PD), clinical attachment level (CAL), healing index (HI), questionnaires will be given to evaluate each of patient perceptions, pain index (PI), and changes in root sensitivity by using visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Good general health.
* No contraindications for periodontal surgery.
* Presence of one localized gingival recession in each side of the maxilla and/or mandible, All recessions will be Class I defects (Miller 1985).
* The cemento-enamel junction (CEJ) is visible in the defective teeth.
* All patients demonstrating good plaque control.
* No previous periodontal surgery in the targeted area.

Exclusion Criteria:

* Smokers.
* pregnant or nursing patients.
* history of malignancy, radiotherapy, or chemotherapy.
* Patients taking medications that affect mucosal healing.
* Patients with allergy to collagen.
* Previous participation in a clinical trial.
* Type-1 diabetes patients.
* Patient who have diseases that affect connective tissue metabolism.

Ages: 18 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-08-25 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Recession depth (REC): (Change in the amount of root coverage) | 1)At baseline, 2) 2 weeks post-surgery, 3) At 1 month post-surgery and 4) 3 months post-surgery.
  from the free gingival margin to the cemento-enamel junction at the mid-buccal aspect. Using University of North Carolina periodontal probe UNC15 (Medesey®-Italy).

SECONDARY OUTCOMES:
change in visible plaque index: | 1) baseline, 2) at 2 weeks postoperative,3) 1 month and 4) 3 month postoperative
  1. Score 0 - No plaque
  2. Score 1 - Separate flecks of plaque at the cervical margin of the tooth
  3. Score 2 - A thin continuous band of plaque at the cervical margin of the tooth
  4. Score 3 - A band of plaque wider then 1mm covering less than 1/3rd of the crown of the tooth
  5. Score 4 - Plaque covering at least 1/3rd but less than 2/3rd of the crown of the tooth
  6. Score 5 - Plaque covering 2/3rd or more of the crown of the tooth
Recession width (RW) | 1) at baseline, 2) at 2 weeks postoperative, 3) at 1 month postoperative, 4) and at 3 months postoperative.
  at the cemento-enamel junction using periodontal probe of University of North Carolina UNC15 (Medesey®-Italy).
Width of keratinized tissue (KT) | 1) baseline, 2) 2 weeks postoperative, 3) 1 month postoperative and 4) 3 months postoperative.
  from the free gingival margin to the mucogingival junction using periodontal probe of University of North Carolina UNC15 (Medesey®-Italy).
Thickness of gingival tissue (GT) | 1) at baseline, and 2) 3 months postoperative.
  with an injection needle and a silicon marker, at the mid-buccal aspect below the gingival margin.
Probing depth (PD) | 1) at baseline, 2) and 3 months postoperative.
  the distance between the gingival margin and the bottom of the pocket measured at the mid-buccal aspect of the tooth using periodontal probe of University of North Carolina UNC15 (Medesey®-Italy).
Clinical attachment level (CAL) | 1) at baseline, 2) at 3 months postoperative.
  distance between the CEJ and the bottom of the pocket measured at the mid-buccal aspect of the tooth using periodontal probe of University of North Carolina UNC15 (Medesey®-Italy).
Healing index | 1) at two weeks following surgery and (2) at one month following surgery.
  score 1 = uneventful healing with no gingival edema, erythema, suppuration, patient discomfort, or flap dehiscence.
  score 2 = uneventful healing with slight gingival edema, erythema, patient discomfort, or flap dehiscence, but no suppuration.
  score 3 = poor wound healing with significant gingival edema, erythema, patient discomfort, flap dehiscence, or any suppuration.
Pain index (PI) | 1) at 2 hours, 2) 24 hours, 3) 48 hours,4) 72 hours following surgery and 5) at 1-week after surgery.
  Using Visual Analogue scale (VAS) (2001 Crichton), Patients will be asked to select among 100 scores (0 indicating no pain at all , 50 indicating average pain, and 100 indicating very painful).
Patient Perceptions | at three months post-surgery.
  Using 100 cm Visual Analogue Scale (VAS)Patients will be asked to select among 100 scores (0 indicating very bad, 50 indicating average, and 100 indicating excellent results).
Change in root sensitivity | 1) at baseline, 2) and at 3 months postoperative.
  Using a 100 cm-visual analog scale (VAS), patients' root sensitivity will be recorded with zero indicating no pain or sensitivity, 50 indicating moderate pain or sensitivity and 100 indicating worst pain or sensitivity possible.

CONTACTS AND LOCATIONS:
Overall Officials: Noor Alhuda Ewaz Ali, DDS, Principal Investigator — MSc student in Periodontics, University of Damascus Dental School; Suleiman Dayoub, DDS MSc PhD, Study Chair — Professor of Periodontics, University of Damascus Dental School; Mohammad Alharissy, DDS MSc PhD, Study Director — Assistant Professor of Periodontics, Academic Staff Member At Wadi International University
Locations (1):
- Department of Periodontics, University of Damascus Dental School, Damascus, Syrian Arab Republic, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim HJ, Chang H, Kim S, Seol YJ, Kim HI. Periodontal biotype modification using a volume-stable collagen matrix and autogenous subepithelial connective tissue graft for the treatment of gingival recession: a case series. J Periodontal Implant Sci. 2018 Dec 27;48(6):395-404. doi: 10.5051/jpis.2018.48.6.395. eCollection 2018 Dec. PMID 30619640
- [Background] Matoh U, Petelin M, Gaspersic R. Split-Mouth Comparison of Coronally Advanced Flap with Connective Tissue Graft or Collagen Matrix for Treatment of Isolated Gingival Recessions. Int J Periodontics Restorative Dent. 2019 May/Jun;39(3):439-446. doi: 10.11607/prd.3562. PMID 30986293
- [Background] Jepsen K, Stefanini M, Sanz M, Zucchelli G, Jepsen S. Long-Term Stability of Root Coverage by Coronally Advanced Flap Procedures. J Periodontol. 2017 Jul;88(7):626-633. doi: 10.1902/jop.2017.160767. Epub 2017 Mar 17. PMID 28304210
- [Background] Lafzi A, Abolfazli N, Faramarzi M, Eyvazi M, Eskandari A, Salehsaber F. Clinical comparison of coronally-advanced flap plus amniotic membrane or subepithelial connective tissue in the treatment of Miller's class I and II gingival recessions: A split-mouth study. J Dent Res Dent Clin Dent Prospects. 2016;10(3):162-8. doi: 10.15171/joddd.2016.026. Epub 2016 Aug 17. PMID 27651882
- [Background] Rasperini G, Acunzo R, Pellegrini G, Pagni G, Tonetti M, Pini Prato GP, Cortellini P. Predictor factors for long-term outcomes stability of coronally advanced flap with or without connective tissue graft in the treatment of single maxillary gingival recessions: 9 years results of a randomized controlled clinical trial. J Clin Periodontol. 2018 Sep;45(9):1107-1117. doi: 10.1111/jcpe.12932. Epub 2018 Aug 20. PMID 29777632
- [Background] Stefanini M, Jepsen K, de Sanctis M, Baldini N, Greven B, Heinz B, Wennstrom J, Cassel B, Vignoletti F, Sanz M, Jepsen S, Zucchelli G. Patient-reported outcomes and aesthetic evaluation of root coverage procedures: a 12-month follow-up of a randomized controlled clinical trial. J Clin Periodontol. 2016 Dec;43(12):1132-1141. doi: 10.1111/jcpe.12626. Epub 2016 Nov 7. PMID 27717210
- [Background] Zucchelli G, Mele M, Mazzotti C, Marzadori M, Montebugnoli L, De Sanctis M. Coronally advanced flap with and without vertical releasing incisions for the treatment of multiple gingival recessions: a comparative controlled randomized clinical trial. J Periodontol. 2009 Jul;80(7):1083-94. doi: 10.1902/jop.2009.090041. PMID 19563288
- [Background] Stefanini M, Zucchelli G, Marzadori M, de Sanctis M. Coronally Advanced Flap with Site-Specific Application of Connective Tissue Graft for the Treatment of Multiple Adjacent Gingival Recessions: A 3-Year Follow-Up Case Series. Int J Periodontics Restorative Dent. 2018 Jan/Feb;38(1):25-33. doi: 10.11607/prd.3438. PMID 29240201
- [Background] Tatakis DN, Trombelli L. Gingival recession treatment: guided tissue regeneration with bioabsorbable membrane versus connective tissue graft. J Periodontol. 2000 Feb;71(2):299-307. doi: 10.1902/jop.2000.71.2.299. PMID 10711621
- [Background] Chambrone L, de Castro Pinto RCN, Chambrone LA. The concepts of evidence-based periodontal plastic surgery: Application of the principles of evidence-based dentistry for the treatment of recession-type defects. Periodontol 2000. 2019 Feb;79(1):81-106. doi: 10.1111/prd.12248. PMID 30892767
- [Background] Jepsen K, Jepsen S, Zucchelli G, Stefanini M, de Sanctis M, Baldini N, Greven B, Heinz B, Wennstrom J, Cassel B, Vignoletti F, Sanz M. Treatment of gingival recession defects with a coronally advanced flap and a xenogeneic collagen matrix: a multicenter randomized clinical trial. J Clin Periodontol. 2013 Jan;40(1):82-9. doi: 10.1111/jcpe.12019. Epub 2012 Oct 10. PMID 23050490
- [Background] de Sanctis M, Zucchelli G. Coronally advanced flap: a modified surgical approach for isolated recession-type defects: three-year results. J Clin Periodontol. 2007 Mar;34(3):262-8. doi: 10.1111/j.1600-051X.2006.01039.x. PMID 17309597